CLINICAL TRIAL: NCT07246460
Title: UPGRADE: Ultrasound and Proteomics for Guselkumab Response Assessment in Crohn's Disease.
Brief Title: Ultrasound and Proteomics for Guselkumab Response Assessment in Crohn's Disease (UPGRADE).
Acronym: UPGRADE
Status: Recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: REB25-0321
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Crohn's Disease of Both Small and Large Intestine
Keywords: Stricture
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Ileal and colonic tissue from endoscopic biopsies Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Inflammatory Ileal Crohn's Disease: Ileal or ileocolonic Crohn's disease patients without fibrostenotic behaviour on endoscopy and diagnostic imaging will receive guselkumab.
  Interventions: Drug: Guselkumab Subcutaneous
- Fibrostenotic Ileal Crohn's disease: Patients with ileal or ileocolonic Crohn's disease with fibrostenotic behaviour on diagnostic imaging will receive guselkumab.
  Interventions: Drug: Guselkumab Subcutaneous

INTERVENTIONS:
Drug: Guselkumab Subcutaneous — Guselkumab will be prescribed by the patient's primary physician according to approved doses by Health Canada for moderate to severe Crohn's disease.
  Dosing includes:
  Induction: 200 mg IV or 400mg sc at Weeks 0, 4, and 8 Maintenance: 100 mg SC every 8 weeks or 200 mg SC every 4 weeks

SUMMARY:
The goal of this observational study is to evaluate the response of guselkumab in adult patients with Crohn's disease (CD) as measured on intestinal ultrasound (IUS), the relative quantities of CD64 in endoscopic tissue biopsies, and the protein signature in the blood of patients with and without therapy response. The main question it aims to answer is:

* What is the proportion of ileal Crohn's disease patients with and without strictures who achieve an intestinal ultrasound response?
* What is the quantity of CD64 in tissue in CD patients at baseline and at week 52 with and without IUS response?
* Are there proteomic signatures in blood of CD patients that respond to GUS?

DETAILED DESCRIPTION:
This is a prospective, single-centre observational study conducted at conducted at the University of Calgary and the University of Alberta. All patients with histologically confirmed distal ileal CD with or without colonic involvement initiating guselkumab (GUS) will be consecutively enrolled. Patients will be sub-divided into the following phenotypes: 1) Stricture: Bowe wall thickness > 3 mm, luminal apposition < 1cm and prestenotic dilation of distal ileum, or 2) Non-Stricture (inflammatory): ileal CD with no evidence of stricture on intestinal ultrasound (IUS) or prior cross-sectional imaging.

Recruited patients providing informed consent will undergo IUS within 14 days of GUS start with blood collection prior to GUS start. Blood collection and IUS will be performed at weeks 0, 12, 24, and 52. Length of visit windows will be within 14 days of study visit due date. Gastroenterologists with bowel sonography expertise will perform standard of care IUS on all consented CD patients meeting inclusion criteria in clinic at baseline, weeks 12, 24, and 52. Colonoscopy will be performed in all patients at baseline and between week 48 and 52 with segmental biopsies for proteomic and CD64 analysis. For tissue CD64 quantification, a single-cell suspension will be obtained using collagenase type 4 and deoxyribonuclease I for enzymatic digestion followed by mechanical dissociation. CD64 will be tagged using the same markers as described for serum, and samples will be submitted to flow cytometry at the local university facility (Calgary or Alberta). Serum will be collected for proteomic analysis at baseline and week 52.

ELIGIBILITY:
Inclusion Criteria:

Male or female, 18 to 80 years old

BWT on IUS > 3.0mm in the ileum and colonic disease permitted.

Patients naïve to guselkumab.

Stricture phenotype - BWT > 3 mm, luminal apposition < 1cm or < 50% of adjacent normal bowel diameter, and prestenotic dilation of distal ileum. Naïve or anastomotic strictures permitted.

Non-stricture phenotype- ileal CD with no evidence of stricture on IUS, computed tomography enterography (CTE), or magnetic resonance enterography (MRE), ever or fistulizing phenotype.

Exclusion Criteria:

Pregnancy

Ileostomy or colostomy

Significant obesity (BMI > 35)

Contraindications to initiating GUS such as active infection.

Active malignancy within five years.

Conditions with fibrosis involving other organs such as lungs, kidneys, brain, or skin.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: University of Calgary IBD Clinic and endoscopy University of Alberta IBD Clinic and endoscopy
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with IUS response in patients with and without Crohn's disease strictures on Guselkumab therapy over 1 year | 52 weeks
  IUS response: decreased bowel wall thickness of > 25%, or > 2.0mm, or > 1.0mm and one colour Doppler signal reduction.
  Transmural remission: Bowel wall thickness < 3mm, colour Doppler signal (modified Limberg grade 0), normal stratification, normal inflammatory fat, and no complications (abscess, phlegmon, fistulas).

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Lu, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared for this study. The study team does not plan to share deidentified individual participant data due to privacy concerns and limitations in consent for data sharing. Compiled results will be disseminated through scientific publications and presentations.

REFERENCES:
- [Result] Kucharzik T, Wilkens R, D'Agostino MA, Maconi G, Le Bars M, Lahaye M, Bravata I, Nazar M, Ni L, Ercole E, Allocca M, Machkova N, de Voogd FAE, Palmela C, Vaughan R, Maaser C; STARDUST Intestinal Ultrasound study group. Early Ultrasound Response and Progressive Transmural Remission After Treatment With Ustekinumab in Crohn's Disease. Clin Gastroenterol Hepatol. 2023 Jan;21(1):153-163.e12. doi: 10.1016/j.cgh.2022.05.055. Epub 2022 Jul 14. PMID 35842121
- [Result] Hart A, Panaccione R, Steinwurz F, Danese S, Hisamatsu T, Cao Q, Ritter T, Seidler U, Olurinde M, Vetter ML, Yee J, Yang Z, Wang Y, Johanns J, Han C, Sahoo A, Terry NA, Sands BE, D'Haens G; GRAVITI Study Group. Efficacy and Safety of Guselkumab Subcutaneous Induction and Maintenance in Participants With Moderately to Severely Active Crohn's Disease: Results From the Phase 3 GRAVITI Study. Gastroenterology. 2025 Aug;169(2):308-325. doi: 10.1053/j.gastro.2025.02.033. Epub 2025 Mar 18. PMID 40113101